CLINICAL TRIAL: NCT07105384
Title: Quantification Tools for a Novel Tau PET Marker in a Rare Neurological Disease: 18F-PI-2620 in Progressive Supranuclear Palsy
Acronym: Quanti-TAU-PET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023-508718-40-00; 2023-508718-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-27; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients suggestive of progressive supranuclear paralysis (Active Comparator): Patients will receive the radiotracer
  Interventions: Combination Product: Radiotracer
- Patients with probable progressive supranuclear palsy (Active Comparator): Patients will receive the radiotracer
  Interventions: Combination Product: Radiotracer
- Control Arm. No pathologies control arm (Active Comparator): Patients will receive the radiotracer
  Interventions: Combination Product: Radiotracer
- Control arm. Patients with parkinson (Active Comparator): Patients will receive the radiotracer
  Interventions: Combination Product: Radiotracer

INTERVENTIONS:
Combination Product: Radiotracer — Patients will receive a brain tau radiotracer

SUMMARY:
The aim of this clinical trial is to explore the potential of novel 2nd generation tau PET radiotracers as biomarkers in cases suggestive of progressive supranuclear palsy (PSP), an atypical form of parkinsonism.

DETAILED DESCRIPTION:
Phase II, uncontrolled, single-center, uncontrolled, drug-controlled clinical trial for the evaluation of a diagnostic test (PI-2620).

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* Patients of both sexes between 40 and 80 years of age.
* The subject must be able to comply with the protocols and procedures necessary for the development of the clinical trial.
* Conformity of the subject or his/her legal representative to voluntarily participate in the study by signing the informed consent form.
* In women, postmenopausal status (one year without menstruation without other medical causes) or negative pregnancy test. Subjects (women and partners of male of childbearing age must accept the commitment to practice sexual abstinence or use highly effective contraceptive methods (hormonal contraceptives that inhibit ovulation, IUD, surgical sterilization) from their inclusion in the study up to one month after the PET scan.

For PSP patients:

* Have a clinical diagnosis of probable soPSP or PSP according to current diagnostic criteria (Höglinger et al. current diagnostic criteria (Höglinger et al. 2017).
* Magnetic resonance imaging (MRI) study that rules out any other relevant neurological pathology. relevant neurological pathology.

For Parkinson patients:

* To have a clinical diagnosis of Parkinson's disease according to established criteria (Postuma et al. 2015).
* Magnetic resonance imaging (MRI) study that rules out any other relevant neurological pathology.

For control patients:

- Absence of clinical history of neuropsychiatric disease.

Exclusion Criteria:

For all patients:

* Diagnosis of relevant central nervous system disease such as:

Huntington's disease, normotensive hydrocephalus, cerebrovascular disease, frontotemporal dementia, Alzheimer's disease, history of major or recurrent traumatic brain injury, history of epilepsy or seizures history of major or recurrent traumatic brain injury, history of epilepsy or seizures(except febrile seizures in childhood without current antiepileptic medication).

* Presence of terminal illness or illnesses that may put the patient's health at risk by participating in the the patient's health by participating in the study or influencing the results of the study or the patient's or on the patient's ability to participate in the study.
* Abuse of alcohol or other legal or illegal drugs (except nicotine).
* Pregnancy.
* Known allergy to PI-2620 or any of the other components of the radiopharmaceutical.
* Any contraindication or impediment to the performance of the PET/CT study with PI-2620.

with PI-2620.

* Subjects who are not capable of understanding and/or complying with the guidelines necessary for the performance of the test (e.g.: interrogation, physical examination, attending the lumbar puncture, attending the visits, etc.) and who do not have responsible accompanying persons who understand and are committed to complying with these guidelines.
* Subjects who do not cooperate or are not capable of complying with the required procedures required for this clinical trial, such as (but not limited to): social disorders that anticipate an evident lack of collaboration, psychopathy, drug or alcohol abuse.
* Subjects or their legal representatives who do not sign the informed consent.
* Legal incapacity and/or circumstances that prevent the subject or his/her legal representatives from understanding the nature, objectives, potential and possible consequences of the trial.
* Treatment with any other investigational drug in the 30 days prior to inclusion.

For PSP patients:

- Diagnosis or suspicion of any parkinsonian syndrome other than PSP such as idiopathic Parkinson's disease, pharmacological parkinsonism, essential tremor, primary dystonias or any other cause that may produce symptoms similar to those of Parkinson's disease.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2028-06-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Differences in uptake levels of PET-PI-2620, a brain tau radiotracer, in participants with a diagnosis suggestive of PSP, probable PSP, Parkinson's and controls without neurological pathology. | Day Zero Visit 1
  The aim of this clinical trial is to explore the potential of novel 2nd generation tau PET radiotracers as biomarkers in cases suggestive of progressive supranuclear palsy (PSP), an atypical form of parkinsonism( Molecular imaging)

SECONDARY OUTCOMES:
Standard optic value ratio(SUVR) from basic core | Day Zero Visit 1
  Ratio of captation compare with healthy captation(ratio)
Standard optic value ratio(SUVR) from cerebral cortex | Day Zero Visit 1
  Ratio of captation in compare of a healthy captation
PI-2620 Captation in compare to demographics as age | Day Zero Visit 1
  PI-2620 captation in relation to age(Captation vs patient age)
PI-2620 Captation in compare to demographics as gender | Day Zero Visit 1
  PI-2620 captation in compare to gender(captation vs male/female)
PI-2620 Captation in compare to demographics as reference Hospital | Day Zero Visit 1
  PI-2620 captation vs reference Hospital
PI-2620 Captation in compare to clinics as PSPRS scale | Day Zero Visit 1, month 6(V2), month12(V3) and month 18(final visit)
  It measures the severity associated with Parkinson's disease(range)
PI-2620 Captation in compare to clinics as PSP-CDS | Day Zero Visit 1, month 6(V2), month12(V3) and month 18(final visit)
  It measures the severity associated with Parkinson's disease(range)
PI-2620 Captation in compare to clinics as Hoen & Yahr classification | Day Zero Visit 1, month 6(V2), month12(V3) and month 18(final visit)
  Disability associated with Parkinson's disease. It helps in describing the progression of the disease(range)
PI-2620 Captation in compare to clinics as Schwab & England daily living activites scale scale | Day Zero Visit 1, month 6(V2), month12(V3) and month 18(final visit)
  Is a method of assessing the capabilities of people with impaired mobility(percentage)
PI-2620 Captation in compare to clinics as Cerebrospinal fluid biomarkers: NfL(neurofilament light chain) | Visit zero, selection visit and last visit(18month visit)
  CSF biomarkers have been found to have the highest diagnostic potential(pg/mL)
PI-2620 Captation in compare to clinics as Cerebrospinal fluid biomarkers: Amyloid beta | Visit zero, selection visit and last visit(18month visit)
  CSF biomarkers have been found to have the highest diagnostic potential(pg/mL)
PI-2620 Captation in compare to clinics as Cerebrospinal fluid biomarkers: tau & 4R-tau | Visit zero, selection visit and last visit(18month visit)
  CSF biomarkers have been found to have the highest diagnostic potential(pg/mL)
PI-2620 Captation in compare to clinics as Cerebrospinal fluid biomarkers: Alfa sinucleyna | Visit zero, selection visit and last visit(18month visit)
  CSF biomarkers have been found to have the highest diagnostic potential(pg/mL)
PI-2620 administration and Patient safety | Day zero(Visit1), day 7(V2), six month(Visit 3), 12 month(V4), and final visit(18 month)
  All the adverse events occurred along the patient participation will be registred(medRA code)
Ophthalmological examination | Month 6 (Visit 3)
  Ophthalmological examination. A standard of care review will be done in order to find abnormalities which may or not had appeared since inclusion. It is a security decission.(Descrption of the abnormality if applies).
Liver function tests | Day zero(Visit 1) and 6 month(Visit 3)
  Blood test where GOT, GGT, GPT, AST, ALT, LDH and Albumin will be tested(g/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Burunat, Barcelona, Barcelona, Spain